CLINICAL TRIAL: NCT02078492
Title: A Prospective Randomized Double-Blind Trial Comparing 3 Doses of Intravenous Ketorolac for Pain Management in the Emergency Department"
Brief Title: A Prospective Randomized Double-Blind Trial Comparing 3 Doses of Intravenous Ketorolac for Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-01-19
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 - 10 mg of Ketorolac (Experimental): Subjects will be administered 10 mg of Ketorolac for pain relief.
  Interventions: Drug: 10 mg of Ketorolac
- Group 2 - 15mg (Experimental): Subjects will be administered 15mg of Ketorolac.
  Interventions: Drug: 15 mg of Ketorolac
- Group 3 - 30mg (Experimental): Subject will receive 30mg of Ketorolac as a part of standard care.
  Interventions: Drug: 30 mg of Ketorolac

INTERVENTIONS:
Drug: 10 mg of Ketorolac — Patients will receive 10 mg of Ketorolac for pain control.
  Other Names: Toradol
  Arms: Group 1 - 10 mg of Ketorolac
Drug: 15 mg of Ketorolac — Patients will receive 15mg of Ketorolac for pain control.
  Other Names: Toradol
  Arms: Group 2 - 15mg
Drug: 30 mg of Ketorolac — Patients will receive 30mg of Ketorolac for pain control.
  Other Names: Toradol
  Arms: Group 3 - 30mg

SUMMARY:
Hypothesis: Intravenous administration of Ketorolac in a dose of 10 mg is as effective in treating severe acute pain in patients presenting to the ED as 15 mg and 30 mg.

DETAILED DESCRIPTION:
Ketorolac tromethamine is a non-steroidal anti-inflammatory drug (NSAID) that is widely used in the Emergency Department (ED) for the treatment of moderate-to-severe pain. Ketorolac is available in both oral and parenteral forms and possess significant analgesic potency. However, ketorolac provides few advantages over other currently available analgesics and its use is limited by a virtue of having an "analgesic ceiling" with the dose being 10mg as well as having a range of severe side effects, of which gastrointestinal hemorrhage is most concerning.The concept of an analgesic ceiling is that doses beyond this value (10mg) do not provide additional analgesia and do contribute to side effects. In spite of this, the majority of research conducted on ketorolac in the ED and recommendations in Tintinalli's Emergency Medicine Textbook advocating for use of three-to-six fold higher dosages.

Hypothesis: Intravenous administration of Ketorolac in a dose of 10 mg is as effective in treating severe acute pain in patients presenting to the ED as 15 mg and 30 mg.

ELIGIBILITY:
Inclusion Criteria:

Severe flank and abdominal pain, severe musculoskeletal pain (traumatic and non-traumatic in origin), headache, dental pain.

Exclusion Criteria:

Age >65, Active Peptic Ulcer disease, Acute Gastrointestinal Hemorrhage, Known Hx of Renal or Hepatic insufficiency, Hx of allergies to NSAIDS.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Motov, MD, Principal Investigator — Attending
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catapano MS. The analgesic efficacy of ketorolac for acute pain. J Emerg Med. 1996 Jan-Feb;14(1):67-75. doi: 10.1016/0736-4679(95)02052-7. PMID 8655940

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 - 10 mg of Ketorolac | Group 2 - 15mg | Group 3 - 30mg
Started | 80 | 80 | 80
Completed | 80 | 80 | 80
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - 10 mg of Ketorolac | Group 2 - 15mg | Group 3 - 30mg | Total
Number analyzed (Participants) | 80 | 80 | 80 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (12.1) | 40.1 (12.1) | 38.8 (11.6) | 40.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 48 | 43 | 132
  Male | 39 | 32 | 37 | 108
Region of Enrollment [Number; unit: participants]
  United States | 80 | 80 | 80 | 240

OUTCOME MEASURES:

1. Primary Outcome: Pain Score at 30 Minutes
Description: Pain score of each group at 30 minutes. The Numeric Rating Pain (NRS) scale was used for the study. The NRS ranges from 0 (no pain) to 10 (very severe pain). A score of 5 is moderate pain. The higher the pain score the higher the pain severity.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: pain score
Arm/Group | Group 1 - 10 mg of Ketorolac | Group 2 - 15mg | Group 3 - 30mg
Number analyzed (Participants) | 80 | 80 | 80
pain score | 5.14 (2.70) | 5.05 (2.56) | 4.81 (2.85)

2. Secondary Outcome: Adverse Effect of Dizziness
Description: the number of study patients who reported having dizziness after administration of medication.
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - 10 mg of Ketorolac | Group 2 - 15mg | Group 3 - 30mg
Number analyzed (Participants) | 80 | 80 | 80
Participants | 14 | 16 | 12

3. Secondary Outcome: Adverse Effect of Nausea
Description: The number of study patients who reported nausea after administration of medication
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - 10 mg of Ketorolac | Group 2 - 15mg | Group 3 - 30mg
Number analyzed (Participants) | 80 | 80 | 80
Participants | 9 | 11 | 8

4. Secondary Outcome: Adverse Effect of Headache
Description: The number of study patients who reported headache after administration of medication
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - 10 mg of Ketorolac | Group 2 - 15mg | Group 3 - 30mg
Number analyzed (Participants) | 80 | 80 | 80
Participants | 8 | 2 | 3
Statistical Analysis 1: Comparison: Group 1 - 10 mg of Ketorolac vs Group 2 - 15mg vs Group 3 - 30mg; The main hypothesis was that there would be equivalence of dose effect across the three groups at every time point, and the primary comparison consisted of the pain assessment at 30 minutes; Test type: Non-Inferiority or Equivalence — We assumed a minimal clinically significant difference (MCSD) of 1.3 between the three ketorolac groups at the 30-minute pain assessment and a standard deviation of 3.0. A power analysis determined that a sample of 78 subjects per group provided at least 80% power to detect an MCSD of at least 1.3 at 30 minutes with α=0.05; p = .783, ANOVA; 2 degrees of freedom

ADVERSE EVENTS:
Arm/Group | Group 1 - 10 mg of Ketorolac | Group 2 - 15mg | Group 3 - 30mg
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes